CLINICAL TRIAL: NCT03287024
Title: Prospective, Multicenter, Single-arm Study to Assess the Safety and Performance of the BeGrow Stent System in Newborns and Infants to Treat Pulmonary Artery Stenosis
Brief Title: BeGrow Study to Treat Pulmonary Artery (PA) Stenosis in Newborns and Infants
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bentley InnoMed GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BNT002BeGrow
Record Dates: First submitted 2017-09-07; First posted 2017-09-19 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Pulmonary Artery Stenosis
MeSH Terms: conditions — Stenosis, Pulmonary Artery

STUDY DESIGN:
Intervention Model Description: Prospective, multi-centre, explorative single-arm study This open-label, non-randomized multi-centre study uses an "umbrella protocol" (Part A and Part B) designed to collect data for performance and safety as well as long-term safety data from pulmonary artery stenosis patients who are treated with the BeGrow stent system to treat the stenosis
  Part A: Safety and Performance (Implantation and Re-dilatation) Part B: Safety on Long-Term Follow-up
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BeGrow Stent System (Experimental): All enrolled subjects will receive the BeGrow Stent System
  Interventions: Device: BeGrow Stent System

INTERVENTIONS:
Device: BeGrow Stent System — All enrolled subjects will undergo primary stenting of the target lesion by placement of the BeGrow Stent System

SUMMARY:
Objective of the study is to assess safety and performance of the BeGrow Stent System for newborns and infants in pulmonary artery stenosis.

DETAILED DESCRIPTION:
The Bentley InnoMed "BeGrow Stent System for Newborns and Infants" is a stent delivery system indicated for intraluminal placement in the pulmonary arteries of newborns and infants for the treatment of Pulmonary Artery Stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Single lesion(s) which can be treated with a 6 mm BeGrow stent (only one stent per lesion allowed).
* Pulmonary artery stenosis - patient must at least have one of the following diseases:

  * Haemodynamically relevant proximal or distal branch pulmonary artery stenosis with a reduction of the vessel diameter when the vessel/patient is large enough to accommodate a stent,
  * Haemodynamically relevant stenosis of the main pulmonary artery segment that results in elevation of the Right Ventricle (RV) pressure, provided that the stent definitely will not compromise a functioning pulmonary valve and will not impinge on the pulmonary artery bifurcation,
  * Any degree of stenosis in patients with single ventricle circulation
  * Critically ill postoperative cardiac patients when it has been determined that branch pulmonary artery stenosis is resulting in a definite haemodynamic compromise in a patient/vessel of any size, particularly if balloon dilatation is unsuccessful
* Signed written informed consent (by parents/legal guardians)
* Lesion can be accessed with a guide wire or balloon catheter
* Age ≤ 24 months and weight ≥ 2 kg
* Adequate stent length available

Exclusion Criteria:

* The following lesions are excluded from treatment with BeGrow stent:

  * Shunt stenosis
  * Valvular and subvalvular pulmonary stenosis
* Patients with known hypersensitivity to the stent material (L605 cobalt-chromium).
* Patients with clinical or biological signs of infection.
* Patients with active endocarditis.
* Patients with known allergy to acetylsalicylic acid, other antiplatelet agents or heparin.
* Presence of other previously implanted stents in the same lesion or in close proximity to stent (direct stent-stent contact).
* Patients with known coagulation disorder.
* Patients where direct stent-stent contact or overlapping cannot be avoided.
* Patients where contact to the vessel wall over the entire stent length cannot be ensured after dilatation (especially in short and thick lesions).
* Patients where the BeGrow stent could protrude freely into adjacent vessels after expansion/dilatation, including the pulmonary arterial bifurcation.
* Implantation of the BeGrow stent in the pulmonary arterial bifurcation.

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Vessel enlargement in mm | after procedure and during follow ups up to 12 Months
  Vessel enlargement will be measured in mm, directly before and after stent implantation by angiography
Incidence of serious adverse events device and procedure related | 12 Months
  Incidence of SAE

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Kretschmar, Prof.Dr.med, Principal Investigator — Kinderspital Zürich, Pädiatrische Kardiologie
Locations (3):
- Medizinische Universität Wien, AKH Wien, Abteilung für Pädiatrische Kardiologie, Vienna, Austria
- University Children's Hospital, Center for Pediatrics - Department of Cardiology, Belgrade, Serbia
- Universitäts-Kinderspital Zürich, Zurich, Switzerland

REFERENCES:
- [Derived] Quandt D, Knirsch W, Michel-Behnke I, Kitzmuller E, Obradovic M, Uhlemann F, Kretschmar O. First-in-man pulmonary artery stenting in children using the Bentley(R) BeGrow stent system for newborns and infants. Int J Cardiol. 2019 Feb 1;276:107-109. doi: 10.1016/j.ijcard.2018.11.029. Epub 2018 Nov 19. PMID 30477928